CLINICAL TRIAL: NCT05820503
Title: Effect of Ultrasound-guided Rectus Abdominis Sheath Block on Analgesia and Agitation During the Awakening Period in Children After Single-port Laparoscopic Inguinal Hernia Repair
Brief Title: Effect of Nerve Block Under Ultrasound on Postoperative Prognosis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-K036
Record Dates: First submitted 2023-03-22; First posted 2023-04-19 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-01

CONDITIONS: Quality of Recovery
Keywords: Nerve block; Hernia in the groin; PAED score; FLACC score
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- R group :Ultrasound-guided lower abdominis rectus sheath block group (Experimental): Under ultrasound guidance, the probe was transversely placed at the lateral level of the umbilicus . Using the in-plane technique, the needle was advanced until the posterior aspect of the rectus muscle was penetrated. No blood and no gas were drawn back; furthermore, a small volume of saline was initially injected to ensure that the needle tip was correctly positioned. When the needle was located between the posterior rectus muscle and posterior sheath, 5ml of 0.25% ropivacaine was injected bilaterally.
  Interventions: Procedure: Ultrasound-guided lower abdominis rectus sheath block
- Control group (No Intervention): Do nothing with it
- Local anesthesia infiltration Group (Experimental): Local anesthesia drugs were injected into the peri-umbilicus cord
  Interventions: Procedure: Local anesthesia infiltration

INTERVENTIONS:
Procedure: Ultrasound-guided lower abdominis rectus sheath block — Under ultrasound guidance, the probe was transversely placed at the lateral level of the umbilicus . Using the in-plane technique, the needle was advanced until the posterior aspect of the rectus muscle was penetrated. No blood and no gas were drawn back; furthermore, a small volume of saline was initially injected to ensure that the needle tip was correctly positioned. When the needle was located between the posterior rectus muscle and posterior sheath, 5ml of 0.25% ropivacaine was injected bilaterally
  Arms: R group :Ultrasound-guided lower abdominis rectus sheath block group
Procedure: Local anesthesia infiltration — Local anesthesia drugs were injected into the peri-umbilicus cord
  Arms: Local anesthesia infiltration Group

SUMMARY:
The goal of this study was to compare the incidence of pain and recovery agitation after single-port laparoscopic inguinal hernia repair in children. The main questions it aims to answer are:

* Reduction of postoperative pain by rectus sheath block compared with local anesthesia infiltration and control group
* A comparison between rectus sheath block and local anesthesia infiltration and control group on the reduction of agitation during postoperative recovery If there is a comparison group: The researchers will compare the ultrasound-guided rectus sheath group with the local anesthesia infiltration group and the control group to look at postoperative pain indicators and the incidence of waking agitation.

DETAILED DESCRIPTION:
Postoperative emergence delirium is a common phenomenon in clinical practice, with an incidence rate of up to 20% to 80%. It has long been a concern and research topic in the medical community. In recent years, with the continuous improvement and updating of anesthesia technology, research on pediatric emergence delirium has become more and more in-depth.

The goal of this study was to compare the incidence of pain and recovery agitation after single-port laparoscopic inguinal hernia repair in children. The main questions it aims to answer are:

* Reduction of postoperative pain by rectus sheath block compared with local anesthesia infiltration and control group
* A comparison between rectus sheath block and local anesthesia infiltration and control group on the reduction of agitation during postoperative recovery If there is a comparison group: The researchers will compare the ultrasound-guided rectus sheath group with the local anesthesia infiltration group and the control group to look at postoperative pain indicators and the incidence of waking agitation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5~12 years old Male and female Single hole inguinal hernia repair surgery should be performed Parents volunteered to participate in the study and signed an informed consent

Exclusion Criteria:

* Preexisting neuropathy Coagulopathy Local skin infection Hepatic, renal, or cardiorespiratory failure Local anesthetic allergy

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Face Legs Activity Cry Consolability (FLACC) score | 0,2, 4, 6, 12, 24, 36, and 48 hours postoperatively
  The Face Legs Activity Cry Consolability (FLACC) scale method is an effective method mainly used for postoperative pain assessment in children . It includes 5 contents: Face, Legs, Activity, Cry and Consolability. Each item is scored on a scale of 0 to 2, with the highest total score being 10. Using the FLACC scale method, doctors need to observe children for 1 to 15 minutes. The pain score is obtained by the medical staff according to the observed children's situation and the content in the quantification table. The total score is obtained by adding up the scores of each content, ranging from 0 to 10. The higher the score, the higher the pain. Doctors can observe children during routine checkups. Touch and change the child's position to determine the child's pain and better assess its body tension and resistance.
Pediatric Anesthesia Emergence Delirium (PAED) scale | Assessments were performed 5 minutes and 10 minutes after awakening, and the highest score was taken
  The PAED scale is a reliable tool for assessing postoperative delirium in children, including 5 scoring items, namely eye contact with caregivers, purposeful activities, cognition of the surrounding environment, and the uneasiness and comfort of children. Each evaluation item can be divided into levels 1 to 5 according to the degree, with 0 to 4 points respectively, and the maximum total score is 20 points. A score of ≥10 on the PAED scale indicates the presence of postoperative delirium, and a score of ≥15 indicates the presence of severe postoperative delirium

SECONDARY OUTCOMES:
Cumulative use of anesthetic drugs during surgery | Perioperative period
  The cumulative use of remifentanil and propofol during the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, Principal Investigator — Ethics Committee of Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No